CLINICAL TRIAL: NCT05122793
Title: "HerzCheck" - Erkennung Und Prävention Einer Frühen Herzinsuffizienz Mittels Telemedizinischer Verfahren in Strukturschwachen Regionen
Brief Title: "HerzCheck" - Detection of Early Heart Failure Using Telemedicine in Structurally Weak Regions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Heart Institute (Other)
Collaborators: medneo GmbH, Germany (Unknown); Medical Statistics, University Medicine of Goettingen (Other); University of Cologne (Other); University Hospital Heidelberg (Other); AOK Nordost (Industry); Herz- und Gefaesszentrum Bad Bevensen (Other)
Responsible Party: Principal Investigator, Sebastian Kelle, Dr. Sebastian Kelle (MD), German Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EA4/204/20
Record Dates: First submitted 2021-10-21; First posted 2021-11-17 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure with Preserved Ejection Fraction
Keywords: Prevention; Heart failure; HFpEF; Asymptomatic; Cardiology; Rural Region; Germany; CMR; Cardiac Magnetic Resonance; HFrEF; Diastolic Dysfunction; Strain; Telemedicine
MeSH Terms: conditions — Heart Failure; Sprains and Strains

STUDY DESIGN:
Intervention Model Description: The present study is a prospective, monocentric, randomised controlled trial with stratification and blinded assessment of the endpoint (Prospective Randomised Open Blinded Endpoint (PROBE) design).
Who Masked: Investigator
Masking Description: The attending physician who examines the patients is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prevention Group (Experimental): In addition to the usual treatment (SoC), the prevention group receives an innovative prevention offer tailored to the severity of the heart failure (telemedical connection via health app as well as additional therapy recommendations).
  Interventions: Behavioral: Prevention offer
- Control Group (No Intervention): The control group receives the current standard treatment according to the valid guidelines (Standard of Care = SoC).

INTERVENTIONS:
Behavioral: Prevention offer — Improvement of outcomes through lifestyle changes and improved health literacy
  Arms: Prevention Group

SUMMARY:
This study is intended to provide a basis for decision-making for the improved medical care of patients with asymptomatic heart failure, especially in structurally weak regions.

DETAILED DESCRIPTION:
The aim of the study is the early detection of asymptomatic heart failure with a quality-assured cardiac screening MRI in the population in structurally weak regions and especially in patients with risk factors for the occurrence of heart failure. The diagnosis is followed by early initiation of appropriate therapeutic measures to improve the prognosis of the affected patients, avoid hospitalisations and save therapy costs, and is combined with recommended measures to minimise risk factors for the development of heart failure. The project includes a prospective, monocentric, randomised controlled clinical trial with blinded assessment of the endpoint (PROBE design). Within the scope of the study, 4,509 patients aged between 40 and 69 years who have characteristic risk factors for the development of heart failure were examined using a mobile cardiac screening MRI in the federal states of Brandenburg and Mecklenburg-Western Pomerania within Germany.

ELIGIBILITY:
Inclusion Criteria:

* Smoking
* Hypercholesterolaemia
* Arterial hypertension
* Obesity
* Chronic diabetes mellitus
* Chronic kidney disease
* Health insurance

Exclusion Criteria:

* Previously diagnosed Heart Failure
* MRI-exclusion criteria

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4509 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
Improved GLS | 12 months
  Improved GLS at after one year compared to baseline.

SECONDARY OUTCOMES:
Body weight in kilograms and body height in meters will be aggregated to report BMI in kg/m^2 | 12 months
  BMI at baseline compared to after one year.
Systolic and diastolic blood pressure in mmHg | 12 months
  blood pressure at baseline compared to after one year.
Heart rate in BPM | 12 months
  heart rate at baseline compared to after one year.
Quality of life questionnaire 1 in Likert scale | 12 months
  Quality of life at after one year compared to baseline. Min. value: 0, max value: 3; higher score: better outcome.
Quality of life questionnaire 2 in Likert scale | 12 months
  Quality of life at after one year compared to baseline. Min. value: 1, max value: 5; higher score: depending on question.
laboratory parameters: Iron, transferrin and creatinine | 12 months
  laboratory parameters in µmol/l at baseline compared to after one year.
laboratory parameters: Sodium, potassium, chloride, total cholesterol, triglycerides, HDL cholesterole, LDL cholesterole, hemoglobin and MCHC | 12 months
  laboratory parameters in mmol/l at baseline compared to after one year.
laboratory parameters: White cells and platelets | 12 months
  laboratory parameters in GPt/l at baseline compared to after one year.
laboratory parameters: MCV | 12 months
  laboratory parameter in fl at baseline compared to after one year.
laboratory parameters: RDW-SD | 12 months
  laboratory parameter in fl at baseline compared to after one year.
laboratory parameter: HbA1c | 12 months
  laboratory parameter in mmol/mol at baseline compared to after one year.
laboratory parameter: red cells | 12 months
  laboratory parameter in TPt/l at baseline compared to after one year.
laboratory parameter: MCH | 12 months
  laboratory parameter in fmol at baseline compared to after one year.
laboratory parameter: hematocrit | 12 months
  laboratory parameter in l/l at baseline compared to after one year.
laboratory parameter: NT-proBNP | 12 months
  laboratory parameter in pmol/l at baseline compared to after one year.
laboratory parameter: transferrin saturation | 12 months
  laboratory parameter in % at baseline compared to after one year.
laboratory parameter: ferritin | 12 months
  laboratory parameter in µg/l at baseline compared to after one year.
hospitalisations of cardiac origin, arrhythmias or death | 12 months
  Appearance of hospitalisations of cardiac origin, arrhythmias or death
Laboratory parameters: urine albumin-creatinine ratio | 12 months
  UACR, calculated from albumin and creatinine in urine in mmol/l at baseline compared to after one year.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Kelle, MD, Principal Investigator — Deutsches Herzzentrum der Charité; Diana Graja, Study Chair — AOK Nordost; Daniel Sievritts, Study Chair — medneo GmbH; Tim Friede, PhD, Study Chair — Medical Statistics, University Medicine of Goettingen; Stephanie Stock, MD, Study Chair — University of Cologne; Norbert Frey, MD, Study Chair — University Hospital Heidelberg; Bjoern Remppis, MD, Study Chair — Herz- und Gefaesszentrum Bad Bevensen
Locations (1):
- Deutsches Herzzentrum der Charité, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
It is not planned to make IPD available to other researchers.

REFERENCES:
- [Background] Biering-Sorensen T, Biering-Sorensen SR, Olsen FJ, Sengelov M, Jorgensen PG, Mogelvang R, Shah AM, Jensen JS. Global Longitudinal Strain by Echocardiography Predicts Long-Term Risk of Cardiovascular Morbidity and Mortality in a Low-Risk General Population: The Copenhagen City Heart Study. Circ Cardiovasc Imaging. 2017 Mar;10(3):e005521. doi: 10.1161/CIRCIMAGING.116.005521. PMID 28264868
- [Background] Liu B, Dardeer AM, Moody WE, Hayer MK, Baig S, Price AM, Leyva F, Edwards NC, Steeds RP. Reference ranges for three-dimensional feature tracking cardiac magnetic resonance: comparison with two-dimensional methodology and relevance of age and gender. Int J Cardiovasc Imaging. 2018 May;34(5):761-775. doi: 10.1007/s10554-017-1277-x. Epub 2017 Nov 27. PMID 29181827
- [Background] Friede T, Kieser M. Sample size recalculation in internal pilot study designs: a review. Biom J. 2006 Aug;48(4):537-55. doi: 10.1002/bimj.200510238. PMID 16972704
- [Background] Huber A, Oldridge N, Benzer W, Saner H, Hofer S. Validation of the German HeartQoL: a short health-related quality of life questionnaire for cardiac patients. Qual Life Res. 2020 Apr;29(4):1093-1105. doi: 10.1007/s11136-019-02384-6. Epub 2019 Dec 12. PMID 31832979
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Rademakers F, Nagel E. Is Global Longitudinal Strain a Superior Parameter for Predicting Outcome After Myocardial Infarction? JACC Cardiovasc Imaging. 2018 Oct;11(10):1458-1460. doi: 10.1016/j.jcmg.2017.11.005. Epub 2017 Dec 13. No abstract available. PMID 29248650
- [Background] Schneider JE, Stojanovic I. Economic evaluation of cardiac magnetic resonance with fast-SENC in the diagnosis and management of early heart failure. Health Econ Rev. 2019 May 23;9(1):13. doi: 10.1186/s13561-019-0229-7. PMID 31123926
- [Background] Tanacli R, Hashemi D, Lapinskas T, Edelmann F, Gebker R, Pedrizzetti G, Schuster A, Nagel E, Pieske B, Dungen HD, Kelle S. Range Variability in CMR Feature Tracking Multilayer Strain across Different Stages of Heart Failure. Sci Rep. 2019 Nov 11;9(1):16478. doi: 10.1038/s41598-019-52683-8. PMID 31712641
- [Background] Unkel S, Amiri M, Benda N, Beyersmann J, Knoerzer D, Kupas K, Langer F, Leverkus F, Loos A, Ose C, Proctor T, Schmoor C, Schwenke C, Skipka G, Unnebrink K, Voss F, Friede T. On estimands and the analysis of adverse events in the presence of varying follow-up times within the benefit assessment of therapies. Pharm Stat. 2019 Mar;18(2):166-183. doi: 10.1002/pst.1915. Epub 2018 Nov 20. PMID 30458579
- [Background] Cosentino F, Grant PJ, Aboyans V, Bailey CJ, Ceriello A, Delgado V, Federici M, Filippatos G, Grobbee DE, Hansen TB, Huikuri HV, Johansson I, Juni P, Lettino M, Marx N, Mellbin LG, Ostgren CJ, Rocca B, Roffi M, Sattar N, Seferovic PM, Sousa-Uva M, Valensi P, Wheeler DC; ESC Scientific Document Group. 2019 ESC Guidelines on diabetes, pre-diabetes, and cardiovascular diseases developed in collaboration with the EASD. Eur Heart J. 2020 Jan 7;41(2):255-323. doi: 10.1093/eurheartj/ehz486. No abstract available. PMID 31497854
- [Background] Chopra VK, Anker SD. Anaemia, iron deficiency and heart failure in 2020: facts and numbers. ESC Heart Fail. 2020 Oct;7(5):2007-2011. doi: 10.1002/ehf2.12797. Epub 2020 Jun 30. PMID 32602663
- [Background] Doeblin P, Hashemi D, Tanacli R, Lapinskas T, Gebker R, Stehning C, Motzkus LA, Blum M, Tahirovic E, Dordevic A, Kraft R, Zamani SM, Pieske B, Edelmann F, Dungen HD, Kelle S. CMR Tissue Characterization in Patients with HFmrEF. J Clin Med. 2019 Nov 5;8(11):1877. doi: 10.3390/jcm8111877. PMID 31694263
- [Background] Fischer F, Gibbons C, Coste J, Valderas JM, Rose M, Leplege A. Measurement invariance and general population reference values of the PROMIS Profile 29 in the UK, France, and Germany. Qual Life Res. 2018 Apr;27(4):999-1014. doi: 10.1007/s11136-018-1785-8. Epub 2018 Jan 19. PMID 29350345
- [Background] Gaggin HK, Januzzi JL Jr. Biomarkers and diagnostics in heart failure. Biochim Biophys Acta. 2013 Dec;1832(12):2442-50. doi: 10.1016/j.bbadis.2012.12.014. Epub 2013 Jan 9. PMID 23313577
- [Background] Pedrizzetti G, Lapinskas T, Tonti G, Stoiber L, Zaliunas R, Gebker R, Pieske B, Kelle S. The Relationship Between EF and Strain Permits a More Accurate Assessment of LV Systolic Function. JACC Cardiovasc Imaging. 2019 Sep;12(9):1893-1895. doi: 10.1016/j.jcmg.2019.03.019. Epub 2019 May 15. No abstract available. PMID 31103586
- [Derived] Kelle S, Nolden AC, Muller ML, Beyer RE, Steen H, Remppis BA, Wieditz J, Kentenich H, Tuit A, Cvetkovic M, Witt UE, Andre F, Schmidt S, Huppertz A, Simic D, Muller D, Shukri A, Issing M, Glardon A, Reber KC, Landmesser U, Frey N, Pieske B, Stock S, Falk V, Friede T, Thiede G. Rationale and design of the HERZCHECK trial: Detection of early heart failure using telemedicine and cardiovascular magnetic resonance in structurally weak regions (NCT05122793). J Cardiovasc Magn Reson. 2025 Summer;27(1):101841. doi: 10.1016/j.jocmr.2025.101841. Epub 2025 Jan 15. PMID 39824461
- See also: Project Website in German language — https://www.herzcheck.org/startseite/